CLINICAL TRIAL: NCT04687813
Title: A Randomized, Double-blind, Placebo-controlled Study of the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Single Doses of FTP 198 in Healthy Volunteers
Brief Title: Safety, Tolerability and Pharmacokinetics of FTP-198 Tablet in Healthy Chinese Volunteers
Acronym: FTP-198
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Haisco Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: FTP198-102
Record Dates: First submitted 2020-12-18; First posted 2020-12-29 (Actual); Last update posted 2023-01-23 (Actual); Status verified 2023-01

CONDITIONS: Healthy
Keywords: FTP-198; IPF; health; phase I

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Who Masked: Participant, Investigator
Masking Description: Double (Participant, Investigator)
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Single Ascending Doses 100mg (Experimental): Drug: FTP-198, single dose 100mg Drug: Placebo, single dose Placebo matched to FTP-198, tablet
  Interventions: Drug: Placebo
- Single Ascending Doses 300mg(food-impact) (Experimental): Drug: FTP-198, single dose 300mg Drug: Placebo, single dose Placebo matched to FTP-198, tablet 2-X: fasting (Period 1) ; 2-Y:Postprandial (Period 1) 2-X:Postprandial (Period 2); 2-Y:fasting (Period 2)
  Interventions: Drug: Placebo
- Single Ascending Doses 400mg (Experimental): Drug: FTP-198, single dose 400mg Drug: Placebo, single dose Placebo matched to FTP-198, tablet
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Placebo — Placebo is a tablet with the same appearance as FTP-198

SUMMARY:
This is a Phase I, single-dose escalation clinical trial for FTP-198 conducted in chinese healthy volunteers. The safety, tolerability, food-impact and pharmacokinetics of FTP-198 tablet in healthy volunteers will be evaluated using a randomized, double-blind, placebo-controlled trial design.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers will be included in Part A or Part B of the study if they satisfy all the following criteria:

  1. Must have given written informed consent before any study-related activities are carried out and must be able to understand the full nature and purpose of the trial, including possible risks and adverse effects;
  2. Adult males and females, 18 to 55 years of age (inclusive) at screening;
  3. Body mass index ≥ 18.0 and ≤ 30.0 kg/m2, with a body weight ≥ 50 kg at screening;
  4. Be nonsmokers (including tobacco, e-cigarettes and marijuana) for at least 1 month prior to first study drug administration;
  5. Medically healthy without clinically significant abnormalities at screening and predose on Day 1, including:

     1. Physical examination without any clinically relevant findings;
     2. Systolic blood pressure in the range of 90 to 160 mmHg and diastolic blood pressure in the range of 50 to 95 mmHg after 5 minutes in supine position;
     3. Heart rate in the range of 50 to 100 bpm after 5 minutes rest in supine position;
     4. Body temperature, between 35.0°C and 37.5°C;
     5. No clinically significant findings in serum chemistry, hematology, coagulation and urinalysis tests as judged by the investigator;
  6. Conventional 12-lead ECG recording in triplicate (the mean of triplicate measurements will be used to determine eligibility at screening and predose on Day 1) consistent with normal cardiac conduction and function, including:

     * Normal sinus rhythm with HR between 50 and 100 bpm, inclusive;
     * QT interval corrected using the Fridericia method (QTcF) between 350 to 450 msec for male subjects and 350 to 470 msec for female subjects, inclusive;
     * QRS duration of < 120 msec;
     * PR interval of ≤ 210 msec;
     * Electrocardiogram morphology consistent with healthy cardiac ventricular conduction and normal rhythm, and with measurement of the QT interval;
     * No family history of short or long QT syndrome;
     * No history of risk factors for torsade de pointes or the diagnosis;
  7. Female participants must:

     1. Be of nonchildbearing potential ie, surgically sterilized (hysterectomy, bilateral salpingectomy, bilateral oophorectomy at least 6 weeks before screening) or postmenopausal (where postmenopausal is defined as no menses for 12 months without an alternative medical cause), or
     2. If of childbearing potential, must have a negative pregnancy test at screening (blood test) and before the first study drug administration (Day -1 urine test). They must agree not to attempt to become pregnant, must not donate ova, and must use a highly effective contraceptive method from signing the consent form until at least 30 days after the last dose of study drug.
  8. Male participants, if not surgically sterilized, must be willing not to donate sperm and, if engaging in sexual intercourse with a female partner who could become pregnant, must be willing to use a condom in addition to having the female partner use a highly effective contraceptive method from signing the consent form until at least 90 days after the last dose of study drug;
  9. Have suitable venous access for blood sampling;
  10. Be willing and able to comply with all study assessments and adhere to the protocol schedule and restrictions.

Exclusion Criteria:

* Healthy volunteers will be excluded from Part A or Part B of the study if there is evidence of any of the following at screening, Day -1 or predose on Day 1:

  1. History or presence of significant cardiovascular, pulmonary, hepatic, renal, hematological, gastrointestinal, endocrine, immunologic, dermatologic or neurological disease, including any acute illness or surgery within the past 3 months determined by the PI to be clinically relevant;
  2. Current infection that requires antibiotic, antifungal, antiparasitic or antiviral medications;
  3. Any history of malignant disease in the last 10 years (excludes surgically resected skin squamous cell or basal cell carcinoma);
  4. Presence of clinically relevant immunosuppression from, but not limited to, immunodeficiency conditions such as common variable hypogammaglobulinemia;
  5. Use of or plans to use systemic immunosuppressive (eg, corticosteroids, methotrexate, azathioprine, cyclosporine) or immunomodulating medications (eg, interferon) during the study or within 4 months prior to the first study drug administration;
  6. Liver function test results (ie, aspartate aminotransferase [AST], alanine aminotransferase [ALT], and gammaglutamyl transferase [GGT]) and total bilirubin must not be elevated more than 1.2-fold above the upper limit of normal (ULN);
  7. Positive test results for active human immunodeficiency virus (HIV), hepatitis B surface antigen (HBsAg) or hepatitis C virus (HCV) antibodies (Abs);
  8. History of active, latent or inadequately treated tuberculosis infection;
  9. Presence or having sequelae of gastrointestinal, liver, kidney, or other conditions known to interfere with the absorption, distribution, metabolism, or excretion of drugs;
  10. Estimated creatinine clearance (CrCl) < 40 mL/min using the Cockcroft-Gault formula or serum creatinine more than 1.5-fold above the ULN;
  11. History of substance abuse or alcohol abuse within 12 months prior to first study drug administration;
  12. Positive drug or alcohol test results;
  13. Use of any prescription or over-the-counter medication (including herbal products, diet aids, and hormone supplements) within 10 days or 5 half-lives of the medication (whichever is longer) prior to the first study drug administration, except occasional use of paracetamol;
  14. Demonstrated clinically significant (required intervention, eg, emergency room visit, epinephrine administration) allergic reactions (eg, food, drug, or atopic reactions, asthmatic episodes) which, in the opinion of the investigator, would interfere with the volunteer's ability to participate in the trial;
  15. Known hypersensitivity to any of the study drug ingredients;
  16. Use of any live vaccinations within 30 days prior to the first study drug administration except for the influenza vaccine;
  17. For women of childbearing potential, a positive serum pregnancy test at screening or a positive urine pregnancy test with confirmatory serum pregnancy test on Day -1;
  18. Donation of blood or plasma within 30 days prior to first study drug administration, or loss of whole blood of more than 500 mL within 30 days prior to randomization, or receipt of a blood transfusion within 1 year of first study drug administration;
  19. Participation in another investigational clinical trial within 60 days prior to the first study drug administration;
  20. Any other condition or prior therapy that in the opinion of the PI would make the volunteer unsuitable for this study, including inability to cooperate fully with the requirements of the study protocol or likelihood of noncompliance with any study requirements;
  21. Is an employee of an investigator or sponsor or an immediate relative of an investigator.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 31 (Actual)
Dates: Start 2020-12-23 (Actual); Primary Completion 2021-02-26 (Actual); Study Completion 2021-03-18 (Actual)

PRIMARY OUTCOMES:
The number and severity of treatment emergent adverse events (TEAEs) | 7 days after the last doses
  To assess the safety and tolerability of single and multiple ascending oral doses of FTP-198 in healthy Chinese subjects

SECONDARY OUTCOMES:
The level of changes of pharmacodynamic biomarkers | within 0.5 hours before administration until 24 hours (single dose) or 48 hours (multiple doses) after administration
  The change-from-baseline values of plasma lysophosphatidic acid (LPA) as PD biomarkers
Cmax | within 0.5 hours before administration until 48 hours after administration
  peak palsma concentration
AUC | within 0.5 hours before administration until 48 hours after administration
  area under the plasma concentration versus time curve
t1/2 | within 0.5 hours before administration until 48 hours after administration
  half-life

CONTACTS AND LOCATIONS:
Locations (1):
- West China Hospital SiChuan University, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No